CLINICAL TRIAL: NCT06856187
Title: A Randomized, Phase II Clinical Study of Second-line Standard Treatment Sequential TAS-102 and Bevacizumab Combined With Local Treatment in Advanced Colorectal Cancer
Brief Title: Second-line Standard Treatment Sequential TAS-102 and Bevacizumab Combined With Local Treatment in Advanced Colorectal Cancer
Acronym: TASBEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Li Wenhua, Department of Medical Oncology, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FudanU.2411307-13
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer (CRC)
Keywords: Colorectal cancer; TAS-102; second-line therapy; maintainance therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Second-line standard therapy sequential TAS-102 and bevacizumab group (Experimental): Second-line induce therapy followed by TAS-102+bevacizumab maintainance therapy combined with local treatment
- Continuous therapy of Standard Treatment Group (Active Comparator): Continuous therapy of standard treatment regimen
  Interventions: Drug: Standard chemotherapy

INTERVENTIONS:
Drug: TAS-102+bevacizumab+local treatment — patients achieve disease control after second-line induction therapy with standard therapy(FOLFOX/FOLFIRI/XELOX/ mXELIRI＋bevacizumab/cetuximab), then achieve TAS-102+bevacizumab+local treatment
Drug: Standard chemotherapy — Standard therapy：FOLFOX/FOLFIRI/XELOX/ mXELIRI±bevacizumab/cetuximab
  Arms: Continuous therapy of Standard Treatment Group

SUMMARY:
This study is a randomized, controlled, open-label, phase II clinical study. This study is designed to evaluate the efficacy and safety of second-line standard treatment sequential TAS-102 and bevacizumab combined with local treatment versus continuous treatment of standard second-line therapy in advanced colorectal cancer.

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label, phase II clinical study. This study is designed to evaluate the efficacy and safety of second-line standard treatment sequential TAS-102 and bevacizumab combined with local treatment versus continuous treatment of standard second-line therapy in advanced colorectal cancer.

In this study, 119 metastatic colorectal cancer patients who reach CR/PR/SD after 3 months second-line treatment will be randomized to receive sequential TAS-102 +bevacizumab combined with local treatment or continuous treatment of previous second-line therapy. The primary endpoint is investigator-assessed time to treatment failure (TTF). Secondary endpoints include ORR, DCR, PFS, OS, safety and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable colorectal adenocarcinoma confirmed by histopathology or cytology;
* Patients who have failed first-line standard therapy and are intended to receive second-line standard therapy;
* At least one measurable lesion according to RECIST 1.1 criteria;
* ECOG Performance Status 0-1;
* Estimated life expectancy ≥3months;
* Adequate major organ function;
* Subjects voluntarily participate in this study, sign the informed consent form, and have good compliance.

Exclusion Criteria:

* Allergy to the investigational drug and/or its excipients;
* Pregnant or lactating women;
* Prior treatment with TAS-102;
* Any CTCAE grade 2 or above toxicity caused by previous treatment that has not yet subsided (excluding alopecia, skin pigmentation, and chemotherapy-induced neurotoxicity);
* Known inherited or acquired bleeding (e.g., coagulopathy) or thrombophilia, as in patients with hemophilia; Current or recent (within 10 days before initiation of study treatment) use of a full-dose oral or injectable anticoagulant or thrombolytic agent for therapeutic purposes (prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed);
* Serious illness, including but not limited to the following:

  1. Patients with other malignant tumors within 5 years before enrollment, except basal cell carcinoma of the skin or carcinoma in situ of the cervix;
  2. Known brain and/or leptomeningeal metastases;
  3. Active infection or fever of unknown origin > 38.5 ° C ;
  4. Poorly controlled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) with a previous history of hypertensive crisis or hypertensive encephalopathy;
  5. Known inherited or acquired bleeding (e.g., coagulopathy)
  6. Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc., occurred within 6 months before the initiation of study treatment;
  7. Severe, unhealed or dehiscence wounds and active ulcers or untreated fractures;
  8. Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure (NYHA Class III or IV) within the last 12 months;
  9. Acute or subacute intestinal obstruction, or chronic inflammatory bowel disease;
  10. There are serious psychological or psychiatric abnormalities that affect the compliance of patients to participate in this clinical study.
* Has undergone major surgical treatment (excluding diagnosis) within 4 weeks before the start of the study or is expected to undergo major surgical treatment during the study period;
* Inability to swallow pills, presence of malabsorption syndrome or any condition affecting gastrointestinal absorption;
* The investigator assessed that it is not appropriate to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | up to approximately 2 years.
  TTF is defined as the time from the date of randomization to the date of the discontinuation of the trial protocol.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to approximately 2 years.
  ORR is defined as the percentage of subjects with complete response (CR) or partial response (PR) by investigator assessment per RECIST criteria, version 1.1.
Disease control rate (DCR) | up to approximately 2 years.
  DCR was defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD).
Progression-free survival (PFS) | up to approximately 2 years.
  PFS is defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.
Overall survival（OS） | up to approximately 2 years.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Adverse Events | up to approximately 2 years.
  AE assessed by NCI-CTCAE v5.0.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) | up to approximately 2 years.
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) during study treatment.
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. More points are considered to have a better outcome.
Progression-free survival(PFS2) | up to approximately 2 years.
  PFS2 is defined as the time from receiving second-line standard therapy until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No